CLINICAL TRIAL: NCT03708991
Title: Effectiveness of PGT-A by Using IVF Versus ICSI for Non-male Factor Infertility: a Pilot Study
Brief Title: Effectiveness of PGT-A: IVF Versus ICSI
Status: Completed | Type: Observational
Sponsor: ART Fertility Clinics LLC (Other)
Responsible Party: Sponsor
Other Study IDs: 1809-ABU-059-ND
Record Dates: First submitted 2018-10-08; First posted 2018-10-17 (Actual); Last update posted 2019-08-07 (Actual); Status verified 2019-08

CONDITIONS: Genetic Condition
Keywords: IVF; ICSI
MeSH Terms: conditions — Genetic Diseases, Inborn

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 9 Months
Biospecimen Retention: Samples With DNA — Trophectoderm biopsies from human blastocysts to determine the ploidy state
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- IVF combined with PGT-A: 5000-10000 motile sperm will be added to the oocyte
  Interventions: Diagnostic Test: IVF combined with PGT-A
- ICSI combined with PGT-A: 1 motile sperm will be injected into the oocyte
  Interventions: Diagnostic Test: ICSI combined with PGT-A

INTERVENTIONS:
Diagnostic Test: IVF combined with PGT-A — trophectoderm biopsy to test the ploidy state of the IVF embryos
  Groups: IVF combined with PGT-A
Diagnostic Test: ICSI combined with PGT-A — trophectoderm biopsy to test the ploidy state of the ICSI embryos
  Groups: ICSI combined with PGT-A

SUMMARY:
The investigators want to investigate if the use of conventional in vitro fertilization (IVF) can generate more euploid embryos as compared to intracytoplasmic sperm injection (ICSI).

To verify this, the investigators will inject half of the oocytes by ICSI and the other half of the oocytes will be inseminated by conventional IVF. The most important aim is to see if IVF is able to generate more euploid embryos.

DETAILED DESCRIPTION:
ICSI is commonly used in pre-implantation genetic testing (PGT) cases to eliminate any risk of sperm DNA contamination. With the switch from cleavage stage biopsy to biopsy of the full (hatching) blastocyst, this potential risk of contamination can be neglected and could allow the use of conventional IVF in PGT cases. Especially in cases of non-male factor infertility, the use of conventional IVF can be applied as a more 'natural' insemination method.

The investigators will perform a pilot study on sibling oocytes including participants with non-male factor infertility and requesting PGT-A (PGT for aneuploidy). If at least 10 cumulus oocyte complexes (COCs) are obtained after oocyte retrieval, half of the oocytes will be subjected to ICSI and the other half to conventional IVF. Preimplantation development is followed by time lapse imaging and blastocysts (day 5-7) fulfilling the biopsy criteria will undergo trophectoderm biopsy to detect the ploidy state and the mitochondrial DNA (mtDNA) copy number.

The main objective is to analyse if the use a more physiological insemination method (IVF) has a beneficial impact on the ploidy state of the blastocyst as compared to ICSI within the same participant. As the embryos will be cultured in a time lapse imaging system, annotations can be made and the differences in maturation rate, fertilization rate and embryo development between both insemination methods can be analysed as secondary outcome parameter. On top of this, the PGT-A outcome will also display the mtDNA copy number which can be compared between IVF and ICSI biopsied sibling blastocyst. Euploid blastocysts will be transferred in subsequent frozen embryo transfer (FET) cycles and give an indication on the clinical outcome between IVF and ICSI.

ELIGIBILITY:
Inclusion Criteria:

* Sperm parameters Sperm concentration before capacitation: >15*106 per ml (WHO) Total motility (PR+NP,%): >40 (WHO) Progressive motility (PR,%):>32 (WHO) Sperm concentration after capacitation: >0.6*106 per ml (not WHO defined) Progressive motility (PR,%):>65 (WHO)
* ≥10 COCs after oocyte retrieval
* BMI ≤30 kg/m2
* Female age 18 to ≤ 40 years
* All ovarian stimulation protocols
* Fresh ejaculates
* Presence or absence of sperm morphology data: as the investigators do not have a diagnostic sperm analysis for all participants, the presence or absence of >4% normal morphology (WHO) will not be taken into account, even with known low (<4%) normal morphology
* Couples requesting PGT-A
* Arab population

Exclusion Criteria:

* If after denudation (ICSI) only 2 mature oocytes are obtained
* If all time lapse spaces are occupied
* If the volume to be added after IVF is insufficient to perform IVF on all needed oocytes
* Presence of >1 *106 per ml round cells in the ejaculate
* If a couple's previous cycle was included in the study

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study population is defined by all couples seeking a fertility treatment due to primary or secondary infertility in IVI RMA Abu Dhabi, for non-male factor infertility in combination with a PGT-A request.
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2018-11-08 (Actual); Primary Completion 2019-04-24 (Actual); Study Completion 2019-08-04 (Actual)

PRIMARY OUTCOMES:
Ploidy state: euploid or aneuploid | 7 days
  trophectoderm biopsy performed between day 5-7 of preimplantation development. These cells will be genetically tested to see if the correct number of chromosomes are present. Euploid embryos can be used for the patient, aneuploid embryos cannot be used for the patient.

SECONDARY OUTCOMES:
mitoscore value: ranges from 10-1500 | 1 day
  the trophectoderm biopsy sample is used to calculate a value indicating the mitochondrial DNA present in the biopt. Lower values are known to be linked to higher implantation rates of the corresponding blastocyst. Higher values have been correlated to aneuploidy.
Maturation rate | 1 day
  The maturation rate is defined as the number of mature oocytes obtained per cumulus complex retrieved for the participants.A mature oocyte is defined as an oocyte that has extruded his fiist polar body and this mature oocyte is ready to be fertilized by the participants sperm.
Morphokinetic development | 7 days
  As embryos are cultured in a time lapse imaging system, pictures will be taken every 20 minutes to follow the development. Each time that the embryos divides, the timing will be registered in the database. Like this, every division made by every embryo is recorded. the time the embryo needs to go from 1 cell to 2 cells, from 2 cells to 3 cells and so on.
Fertilization rate | 1 day
  Fertilization is calculated on all mature oocytes or on all complexes obtained after oocyte retrieval. The fertilization rate is assessed by the presence of a male and a female pronucleus 16-20 hours post fertilization. If the oocyte is fertilized, the outcome is positive, if the oocyte is not fertilized, the outcome is negative.
Embryo development up to day 3 | 3 days
  For all normally fertilized oocytes the further development will be assessed as the embryos are cultured in a time lapse system. This system takes pictures of the embryos every 20 minutes which shows the development of the embryo like a movie: every time that a cell divides, the hour at which it divides will be registered in the time lapse system. For each cell division, specific time frames have been described that link the embryo to develop into a blastocyst or that increases the chance of implantation. The embryo will be evaluated on day 3 and will receive an embryo score that is based on the number of cells, the appearance of the cells, fragmentation and embryo dysmorphisms. These will divide the embryo quality into 4 categories with category 1 being the highest quality and category 4 being the lowest quality. The more fragmentation and the higher the degree of dysmorphisms, the more the quality will shift to category 4.
Blastulation rate | 7 days
  A blastocyst is an embryo in which a cavity is visible on day 5 of the embryo development. If the cavity is present the outcome is positive, if the cavity is absent, the outcome is negative The complete process in which the development of one embryo is followed from the day of injection up until day 7 is called the preimplantation development
Embryo development up to day 5 | 7 days
  On day 5 of development, a score is given to every embryo. This is based on the presence or absence of a cavity, the number of cells and how tight the cells are packed. The more cells, the higher the grade, if less cells are present, the grade is lower. Based on these parameters, a final grade is calculated (3 grades) with grade 1 being the highest score.
Pregnancy outcome | 3 months
  pregnancy outcomes from the frozen embryo transfers: blood samples will be taken and the level of beta-hCG will be measured to define a pregnancy or no pregnancy. A pregnancy is defined as the best oucome. In case a pregnancy is obtained, the patient will come for an ultrasound scan between week 7-12 to checke the presence of a gestational sac and the presence of a fetal heart beat. The presence of a fetal heart beat is defined as a positive outcome, the absence is defined as a negative outcome.

OTHER OUTCOMES:
sperm concentration | 1 day
  concentration will be analysed under a microscope in a Makler or Neubauer counting chamber that allows you to define the concentration of that specific sample: depending on the number of sperm cells counted per row or square in the chamber, the concentration can be calculated.
  Concentration will start at 15 million per milliliter in the original sperm and may be as high as 500 million per milliliter.
sperm motility | 1 day
  The motility of the sperm will be analysed under a microscope in a Makler or Neubauer counting chamber that allows you to count the four different types of motility present in a sample.
  Sperm motility is defined as the number of sperm cells that are able to progress on their own and is expressed as a percentage: the higher the percentage, the better the value is.
Controlled ovarian stimulation: dosage | 2 weeks
  In order to stimulate multiple follicular development, patients will be stimulated with fixed doses of hormones. The total dosage of hormones used will be registered.
Controlled ovarian stimulation: days of stimulation | 2 weeks
  In order to stimulate multiple follicular development, patients will be stimulated with fixed doses of hormones. Once the follicular development is optimal (based on the number of follicles and the corresponding hormonal values) the patient can be triggered for final oocyte maturation. The total number of days needed during this stimulation will be registered.
Controlled ovarian stimulation: hormonal profile | 2 weeks
  During the stimulation, the hormonal profile of every patient will be measured (estrogens, luteinizing hormone, progesterone): these blood values will be compared to the number of follicles that are measured in the participants and the combination of the three blood values should correspond to the sizes and numbers of follicles measured in the participants,
Controlled ovarian stimulation: type of trigger | 2 weeks
  Once all follicles have reached the optimal size, the participants will be triggered for final oocyte maturation. The type of trigger that is administered will be recorded.
Controlled ovarian stimulation: measurement of follicles | 2 weeks
  During the stimulation, the follicles present in the participants will grow steadily and the size of the follicles will be measured to ensure a good development (in combination with the hormonal profile). These follicles will be measured by vaginal echography.

CONTACTS AND LOCATIONS:
Overall Officials: Neelke De Munck, PhD, Principal Investigator — IVIRMA Abu Dhabi
Locations (1):
- IVI RMA Abu Dhabi, Abu Dhabi, United Arab Emirates

IPD SHARING:
Plan to Share IPD: Undecided
Information regarding primary and secondary outcome measures will only be shared with researchers from the clinic, involved in the study.

REFERENCES:
- [Background] Li Z, Wang AY, Bowman M, Hammarberg K, Farquhar C, Johnson L, Safi N, Sullivan EA. ICSI does not increase the cumulative live birth rate in non-male factor infertility. Hum Reprod. 2018 Jul 1;33(7):1322-1330. doi: 10.1093/humrep/dey118. PMID 29897449
- [Result] Sahin L, Bozkurt M, Sahin H, Gurel A, Caliskan E. To compare aneuploidy rates between ICSI and IVF Cases. Niger J Clin Pract. 2017 Jun;20(6):652-658. doi: 10.4103/1119-3077.208959. PMID 28656917
- [Result] Feldman B, Aizer A, Brengauz M, Dotan K, Levron J, Schiff E, Orvieto R. Pre-implantation genetic diagnosis-should we use ICSI for all? J Assist Reprod Genet. 2017 Sep;34(9):1179-1183. doi: 10.1007/s10815-017-0966-7. Epub 2017 Jun 13. PMID 28612309
- [Derived] De Munck N, El Khatib I, Abdala A, El-Damen A, Bayram A, Arnanz A, Melado L, Lawrenz B, Fatemi HM. Intracytoplasmic sperm injection is not superior to conventional IVF in couples with non-male factor infertility and preimplantation genetic testing for aneuploidies (PGT-A). Hum Reprod. 2020 Feb 29;35(2):317-327. doi: 10.1093/humrep/deaa002. PMID 32086522